CLINICAL TRIAL: NCT04323163
Title: Yoga, Aerobic and Stretching Exercise Effects on Neurocognitive Performance: A Randomized Controlled Trial
Brief Title: Yoga, Aerobic and Stretching Exercise Effects on Neurocognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Principal Investigator, Neha P. Gothe, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20714
Record Dates: First submitted 2020-03-18; First posted 2020-03-26 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Aging; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga Group (Experimental): Participants will be led through a beginner yoga course taught by a certified yoga instructor. Classes will meet three times a week for 60 minutes over the 6 month study duration. Sessions will focus on yoga postures, breathing, and meditative practices and may utilize mats, blocks, belts, and blankets.
  Interventions: Behavioral: Physical Activity
- Aerobic Group (Experimental): Trained exercise instructors will lead participants through an aerobic group exercise class. Sessions will begin with a 15-20 minute aerobics class and increase in duration over the 6 months capping off at 40-minutes per session. The prescribed intensity will be 50-60% of the maximum heart rate reserve for weeks one to six and 60-75% for the remainder of the program.
  Interventions: Behavioral: Physical Activity
- Stretching Toning Group (Active Comparator): Participants randomized to this group will meet three times a week for an hour-long structured group exercise session. This group will perform stretching and toning exercises using resistance bands, balance disks, and exercise mats.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — 3 sessions per week, 60 minutes per session for 6 months

SUMMARY:
The investigators propose to conduct a 6-month 3-arm randomized controlled exercise trial among older adults to compare the efficacy of yoga with aerobic exercise and stretching-toning exercises on cognitive function, brain structure and function, cardiorespiratory fitness, functional fitness, and inflammatory and molecular markers. Using a single-blind, three arm randomized control trial, 168 older adults ages 55-79 will be assigned to either: a Hatha yoga group, an aerobic exercise group or an active stretching and toning control group. The groups will engage in hour-long group exercise sessions 3x/week. A comprehensive neurocognitive test battery, brain imaging, cardiovascular fitness test, and a blood draw will take place at baseline; end of the 6-month intervention, and at 12-month follow-up.

The proposed work will examine the relationship between yoga training and improved cognitive functioning as well as identify neurobiological correlates as potential mechanisms of action through which yoga training exerts its effect on cognitive function.

COVID-19 Precautions: Due to COVID-19, all exercise sessions will be conducted live via Zoom video-conferencing such that 1/3rd of the participants in each group will exercise in person with the research staff at UIUC campus once a week while the remaining 2/3rd will tune in via Zoom

ELIGIBILITY:
Inclusion Criteria:

* 55-79 years of age at study enrollment
* TICS-M score of 32 or higher
* No current or past diagnosis of mild cognitive impairment or dementias
* Low-active (≤ 2 days of 30 minutes of structured exercise/week)
* Physician's consent to participate in VO2max testing and the exercise program
* Ambulatory
* Absence of health conditions that may be exacerbated by exercise
* Good or corrected vision and hearing
* No MRI contraindications (e.g. metal or implanted devices in the body)
* Right-handed
* Intention to remain in the Champaign-Urbana area over the study duration

Exclusion Criteria:

* Below 55 or above 79 years of age at study enrollment
* TICS-M score of 31 or lower
* Current or past diagnosis of mild cognitive impairment or dementias
* High-active (3 or more days of 30 minutes of structured exercise/week)
* Physician's non-consent to participate in VO2max testing and the exercise program
* Non-ambulatory (use of wheelchairs or walkers)
* Presence of health conditions that may be exacerbated by exercise
* Poor vision and hearing
* MRI contraindications (e.g. metal or implanted devices in the body)
* Left-handed
* Plans to travel outside of Champaign-Urbana area during the study

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | Baseline, 6 months, 12 months
  A comprehensive neuropsychological battery (part of the NIH toolbox) will be used that assesses different domains of cognitive function, including working memory, attention and executive function.

SECONDARY OUTCOMES:
Change in brain structure | Baseline, 6 months, 12 months
  MRI will be used to measure brain volume.
Change in brain function | Baseline, 6 months, 12 months
  Functional MRI will be used to measure changes in brain activity during resting state.

OTHER OUTCOMES:
Changes in physiological biomarkers | Baseline, 6 months, 12 months
  Brain-derived neurotrophic factor (BDNF) will be assessed through a blood serum analysis at each timepoint.
Changes in cardiovascular fitness | Baseline, 6 months, 12 months
  The mediating role of cardiorespiratory fitness will be assessed by using a treadmill based graded exercise test designed to measure peak VO2 capacity

CONTACTS AND LOCATIONS:
Overall Officials: Neha P Gothe, MA, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Given the pilot nature of the study and limited study outcomes, we do not expect to receive requests from other researchers to analyze our datasets. The primary and secondary outcomes and exploratory biomarker data will be published by the Investigative team.

REFERENCES:
- [Derived] Gothe NP, Erlenbach E, Garcia V, Malani R, Voss S, Camacho PB, McAuley E, Burd N, Sutton BP, Damoiseaux JS. Yoga, aerobic and stretching exercise effects on neurocognition: Randomized controlled trial protocol. Contemp Clin Trials. 2023 Aug;131:107240. doi: 10.1016/j.cct.2023.107240. Epub 2023 May 25. PMID 37244365